CLINICAL TRIAL: NCT04559945
Title: The LEADLESS II IDE Study (Phase II): A Safety and Effectiveness Trial for a Leadless Pacemaker System
Brief Title: The LEADLESS II IDE Study for the Aveir VR Leadless Pacemaker System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10226
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Cardiac Rhythm Disorder; Bradycardia
Keywords: Bradycardia; Pacemaker; Leadless
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aveir VR Leadless Pacemaker (Experimental): VVIR pacing
  Interventions: Device: Aveir VR Leadless Pacemaker System

INTERVENTIONS:
Device: Aveir VR Leadless Pacemaker System — Patients will undergo an attempted leadless pacemaker implant

SUMMARY:
prospective, non-randomized, multi-center, international clinical study is designed to confirm the safety and effectiveness of the Aveir LP System in a subject population indicated for a VVI(R) pacemaker.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have one of the clinical indications before device implant in adherence with Medicare, ACC/AHA/HRS/ESC single chamber pacing guidelines including:

   * Chronic and/or permanent atrial fibrillation with 2° or 3° AV or bifascicular bundle branch block (BBB block), including slow ventricular rates (with or without medication) associated with atrial fibrillation; or
   * Normal sinus rhythm with 2° or 3° AV or BBB block and a low level of physical activity or short expected lifespan (but at least one year); or
   * Sinus bradycardia with infrequent pauses or unexplained syncope with EP findings; and
2. Subject is ≥18 years of age; and
3. Subject has a life expectancy of at least one year; and
4. Subject is not enrolled in another clinical investigation; and
5. Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams; and
6. Subject has been informed of the nature of the study, agrees to its provisions and has provided a signed written informed consent, approved by the IRB/EC; and
7. Subject is not pregnant and does not plan to get pregnant during the course of the study.

Exclusion Criteria:

1. Subject has known pacemaker syndrome, has retrograde VA conduction, or suffers a drop in arterial blood pressure with the onset of ventricular pacing; or
2. Subject is allergic or hypersensitive to < 1 mg of dexamethasone sodium phosphate (DSP);
3. Subject has a mechanical tricuspid valve prosthesis; or
4. Subject has a pre-existing endocardial pacing or defibrillation leads; or
5. Subject has current implantation of either conventional or subcutaneous implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device; or
6. Subject has an implanted vena cava filter; or
7. Subject has evidence of thrombosis in one of the veins used for access during the procedure; or
8. Subject had recent cardiovascular or peripheral vascular surgery within 30 days of enrollment; or
9. Subject has an implanted leadless cardiac pacemaker or
10. Subject is implanted with an electrically-active implantable medical device with stimulation capabilities (such as neurological or cardiac stimulators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Complication-Free Rate | 6 weeks
Complication-Free Rate | 12 months
Pacing thresholds and R-wave amplitudes within the therapeutic range | 6 Weeks
Pacing thresholds and R-wave amplitudes within the therapeutic range | 12 months

SECONDARY OUTCOMES:
Appropriate and proportional rate response during graded exercise testing | 3 month follow up
Survival Rate of Patients implanted with the Nanostim Leadless Pacemaker | 2 years

CONTACTS AND LOCATIONS:
Locations (53):
- United States (38):
  - University Hospital - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - The Heart Center PC, Huntsville, Alabama
  - Honor Health, Scottsdale, Arizona
  - University of Southern California, Long Beach, California
  - Premier Cardiology Inc, Newport Beach, California
  - Huntington Memorial Hospital, Pasadena, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Naples Heart Rhythm Specialists PA, Naples, Florida
  - Orlando Health, Orlando, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - St. Elizabeth Medical Center - South Unit, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Ascension St. John Hospital, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Jersey Shore University Medical Center, Ocean Township, New Jersey
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Cardiac Arrhythmia & Pacemaker Center, Roslyn, New York
  - Cone Health Medical Group HeartCare, Greensboro, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Memorial Hermann Hospital, The Woodlands, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - HSC, Eastern Health, St. John's, Newfoundland and Labrador
  - Kinsgston General Hospital, Kingston, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Institut de Cardiologie de Quebec (Hospital Laval), Québec, Quebec
- Na Homolce Hospital, Prague, Czechia
- France (3):
  - CHRU Albert Michallon, Grenoble
  - Hopital d'adulte de la Timone, Marseille
  - CHRU Hopital de Pontchaillou, Rennes
- Centro Cardiologico Monzino, Milan, Italy
- Netherlands (2):
  - Amsterdam Academic Medical Centre (AMC), Amsterdam
  - Isala - ZWolle, Zwolle
- Hospital Universitario Infanta Cristina, Badajoz, Spain
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Exner DV, Doshi R, Tomassoni G, Bunch TJ, Friedman P, Estes NAM, Neuzil P, de la Concha JF, Cantillon DJ; LEADLESS II Investigators. 1-Year Outcomes of a Leadless Ventricular Pacemaker: The LEADLESS II (Phase 2) Trial. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 2):1187-1189. doi: 10.1016/j.jacep.2023.01.031. Epub 2023 Mar 22. No abstract available. PMID 36951813